CLINICAL TRIAL: NCT06171386
Title: Microneedling vs Dermabrasion for Early Facial Scar Resurfacing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00102716
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Scar
Keywords: Dermabrasion; Microneedling; Surgical scars
MeSH Terms: conditions — Cicatrix | interventions — Percutaneous Collagen Induction; Dermabrasion

STUDY DESIGN:
Intervention Model Description: Patients will be invited to participate in the study through the clinic setting - aim to have around 30 patient volunteers. Of the 30 patients, 15 will be randomized to receive microneedling, and 15 will receive dermabrasion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microneedling (Active Comparator): microneedling is a form of collagen induction therapy, often used in conjunction with platelet-rich plasma or hyaluronic acid - Patients will receive two treatments, once at 6-8 weeks following facial surgery, and the second at 12-16 weeks following facial surgery
  Interventions: Procedure: Microneedling
- dermabrasion (Active Comparator): dermabrasion is a technique that improves the skin structure, quality, and appearance of scars through collagen remodeling and reepithelization - Patients will receive the standard of care treatment 6-10 weeks following facial surgery
  Interventions: Procedure: Dermabrasion

INTERVENTIONS:
Procedure: Microneedling — a form of collagen induction therapy
  Arms: microneedling
Procedure: Dermabrasion — a technique that improves the skin structure, quality, and appearance of scars through collagen remodeling and reepithelization
  Arms: dermabrasion

SUMMARY:
This study aims to determine whether microneedling or dermabrasion in the early post-operative period is superior in improving the appearance of surgical scars on the face.

DETAILED DESCRIPTION:
Microneedling and dermabrasion are two common modalities that may be performed in-office to treat surgical scars.

Microneedling is a form of collagen induction therapy, often used in conjunction with platelet-rich plasma or hyaluronic acid.

Dermabrasion is a technique that improves the skin structure, quality, and appearance of scars through collagen remodeling and reepithelization.

To determine which modality is most effective, a prospective study; randomizing a volunteer sample of adult patients with new surgical vertical forehead scars will receive either dermabrasion or microneedling in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer adult patients will be identified by visiting the Facial Plastics and Reconstructive Surgery Clinic at Atrium Health Wake Forest Baptist.
* Patients will be 18 years old+ and have a vertical surgical scar in the superior 1/3 of the face (trichion to glabella).
* Patients will enroll in the clinic research registry and indicate an interest in being involved in the study.

Exclusion Criteria:

* Patients who rate Types 4-6 on the Fitzpatrick scale will be excluded due to risk of poor outcome from dermabrasion.
* There are no other planned exclusion criteria. Patients will not be excluded on the basis of gender, race/ethnicity, or age, provided that they meet the described inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Vancouver Scar Scale Scores | Month 7
  Four characteristics of the scar are assessed. These are: vascularity, height, pliability, and pigmentation. Each characteristic is given a score, which are added together to give an overall score between 0 and 13 - lower scores denoting normal skin
Change in Patient and Observer Scar Assessment Scale Scores | Month 7
  Items and total scale scores for the patient and observer: Each item on both scales has a score of 1 to 10. The lowest score is 1 and corresponds to the normal skin situation. The total score of both scales can be calculated simply by adding the scores of each of the six items. The total score will range from 6 to 60 - lower scores denoting normal skin
Change in Global Aesthetic Improvement Scale Scores | Month 7
  5-point scale wherein 2 = much improved (marked improvement in appearance), 1 = improved (improvement in appearance but a touch-up or re-treatment is indicated - lower scores denoting normal skin

SECONDARY OUTCOMES:
Patient perceived benefit | At time of procedure (pain scale); at 6 months (yes/no)
  At the time of intervention, patients will be asked to rank pain of procedure on a scale of 1-10 (1: minimal discomfort, 10: severe pain). At 6 months, they will also give a yes/no response as to whether they would undergo the study protocol (procedure) again.

CONTACTS AND LOCATIONS:
Overall Officials: Candace M Water, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
photo documentation, de-identified, for review of scar appearance after treatment
Time Frame: Data will become available after all data collection is complete in order to perform independent blinded analysis of scars at all time points.
Access Criteria: Researchers on the study protocol involved in scar assessment